CLINICAL TRIAL: NCT00745914
Title: A Randomized Placebo-Controlled Study to Evaluate the Efficacy of Peroxisome Proliferator-Activated Receptor-gamma (PPAR-gamma) Agonist in Inducing Carotid Atherosclerotic Plaque Regression in Diabetic End-Stage Renal Disease Patients
Brief Title: Peroxisome Proliferator-Activated Receptor-gamma (PPAR-gamma) Agonist in Diabetic End-Stage Renal Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Angela Yee-Moon Wang, Dr, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A111-103
Record Dates: First submitted 2008-09-01; First posted 2008-09-03 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Endstage Renal Disease; Diabetes
Keywords: PPAR-gamma, diabetic, kidney disease, atherosclerosis
MeSH Terms: conditions — Diabetes Mellitus; Kidney Diseases; Atherosclerosis | interventions — Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Pioglitazone drug 15mg daily for 3 months then 30mg for 9 months (Peroxisome Proliferator-Activated Receptor-gamma agonist)
  Interventions: Drug: Pioglitazone
- 2 (Placebo Comparator): placebo comparator drug 15mg daily for 3months, then 30mg for 9 months
  Interventions: Drug: Placebo comparator

INTERVENTIONS:
Drug: Pioglitazone — oral Pioglitazone 15mg daily for 12 weeks, then 30mg daily for 36 weeks
  Other Names: Actos
  Arms: 1
Drug: Placebo comparator — Placebo comparator
  Other Names: Placebo
  Arms: 2

SUMMARY:
To test the hypothesis that PPAR-gamma agonist, rosiglitazone, induces carotid plaque regression in diabetic ESRD patients on maintenance PD via its anti-inflammatory property.

DETAILED DESCRIPTION:
End-stage renal disease (ESRD) patients are at an increased risk of accelerated atherosclerosis and cardiovascular morbidity and mortality. Non-traditional risk factors such as inflammation and insulin resistance have important contributions to accelerated atherosclerosis in ESRD patients receiving long-term peritoneal dialysis (PD). The peroxisome proliferator-activated receptor-g (PPAR-g) is a member of the nuclear receptor family of ligand-dependent transcription factors. Activation of the PPAR-g has been shown in both clinical and experimental studies to have anti-inflammatory and anti-atherosclerotic properties other than insulin-sensitizing effects. Recent study also showed that PPAR-g agonists reduce plaque inflammation by inhibiting the activation of proinflammatory genes responsible for plaque development and growth. Hence, this study aims to examine the effects of PPAR-g activation on the progression of carotid plaque in diabetic ESRD patients receiving long-term PD using high-resolution magnetic resonance imaging (MRI).

ELIGIBILITY:
Inclusion Criteria:

* Diabetic ESRD patients receiving long-term PD treatment, with carotid plaque (defined as focal intima-media thickening >1mm) present on screening ultrasonography
* Patients who provide informed consent for the study

Exclusion Criteria:

* Patients with systemic inflammatory disease such as systemic lupus erythematosus
* Patients with chronic liver disease or cirrhosis
* Patients with current active malignancy
* Patients with chronic rheumatic heart disease or congenital heart disease
* Patients with poor general condition
* Patients with plan for living related kidney transplant within coming 1 year
* Patients with pre-existing class III/IV heart failure,
* Patients with recurrent hypoglycemia
* Patients already on glitazone treatment
* Female patients with pregnancy
* Patients with contraindications for MRI examination including those with pacemaker or metallic implant.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-09; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in carotid plaque volume | 12 months

SECONDARY OUTCOMES:
Change in inflammatory markers include C-reactive protein, interleukin-6, adiponectin, metalloproteinases | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Angela YM Wang, MD, FRCP, Principal Investigator — Queen Mary Hospital, University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Queen Mary Hospital and Tung Wah Hospital, Hong Kong, Hong Kong
  - Queen Mary Hospital, Tung Wah Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: No